CLINICAL TRIAL: NCT03875365
Title: Institutional Outcome Data From Per-oral Plication of the Esophagus (POPE)
Brief Title: Institutional Outcome Data From Per-oral Plication of the Esophagus
Status: Terminated | Type: Observational
Why Stopped: PI left the institution before enrollment was complete.
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 18-007834
Record Dates: First submitted 2019-02-18; First posted 2019-03-14 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-03

CONDITIONS: Achalasia
Keywords: POPE
MeSH Terms: conditions — Esophageal Achalasia | interventions — 1-palmitoyl-2-oleoylphosphatidylethanolamine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- POPE Patients: Patients who underwent POPE for end-stage achalasia, a sigmoid esophagus, or a redundant conduit that has been used to replace the esophagus.
  Interventions: Procedure: POPE

INTERVENTIONS:
Procedure: POPE — Patients who have undergone Per-oral Plication of the Esophagus (POPE) procedure.

SUMMARY:
Researchers are reviewing and analyzing surgical and clinical outcomes of subjects who underwent POPE for end-stage achalasia, a sigmoid esophagus, or a redundant conduit that has been used to replace the esophagus. This data will help researchers determine the safety and efficacy of a novel minimally invasive treatment compared to invasive surgery.

DETAILED DESCRIPTION:
Researchers will be collecting electronic medical data for subjects who have already undergone Per-oral Plication of the Esophagus (POPE) procedure. Subject characteristics, radiographic documentation, videos, procedural details, and subject reported outcomes would be collected. This data will be used for review and analysis to answer questions aimed in this study. Data collected from this study will be entered into a database that will be maintained for future research.

ELIGIBILITY:
Inclusion Criteria:

* Adults > 18 years of age
* Patients who have already undergone Per-oral Plication of the Esophagus (POPE) procedure

Exclusion Criteria:

* Patients <18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have already undergone Per-oral Plication of the Esophagus (POPE) procedure for end-stage achalasia, a sigmoid esophagus, or a redundant conduit that has been used to replace the esophagus.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-01-19 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 01/01/2017-9/17/2018
  Evaluate safety by assessment of adverse events of the novel minimally invasive treatment compared to invasive surgery.
Patient Reported Outcomes using the CONDUIT patient questionnaire. | 01/01/2017-9/17/2018
  Evaluate efficacy by reviewing patient reported outcomes of the novel minimally invasive treatment compared to invasive surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Shanda Blackmon, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials